CLINICAL TRIAL: NCT01280773
Title: Department of Critical Care Medicine, Nanjing Zhong-Da Hospital, Southeast University School of Medicine, China; Department of Critical Care Medicine St. Michaels's Hospital, University of Toronto, Canada
Brief Title: Effect of NAVA on Weaning Duration in Difficult to Wean Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ling Liu (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor-Investigator, Ling Liu, professor, Southeast University, China
Organization: Southeast University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 437129518
Record Dates: First submitted 2010-12-28; First posted 2011-01-21 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Weaning
Keywords: weaning, mechanical ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PSV weaning (No Intervention): Patinens in the PSV group will be weaned using PSV mode.
- NAVA weaning (Experimental): Patients in NAVA group will eb weaned using NAVA mode.
  Interventions: Device: NAVA

INTERVENTIONS:
Device: NAVA — Neurally adjusted ventilatory assist (NAVA) was delivered by a SVi ventilator. NAVA utilizes EAdi, a reflection of the neural respiratory output to diaphragm, as its primary source to trigger and cycle-off assist in synchrony with neural inspiratory efforts.
  Arms: NAVA weaning

SUMMARY:
It has been showed that over assist and patient ventilator asynchrony often occur in mechanical ventilated patients, especially in patients who failed weaning, which are associated with a prolonged duration of mechanical ventilation.Neurally adjusted ventilatory assist (NAVA) improves patient-ventilator synchrony, prevents excessive assist induced diaphragm inactivation. So the aim of this study was to detect that whether NAVA compared with PSV has the ability to reduce the duration of weaning in difficult to wean patients.

DETAILED DESCRIPTION:
Intubated patients who were deemed ready for weaning by the clinical team but failed the first spontaneous breathing trials (SBT) or weaning were screened for eligibility. After enrollment, nasogastric tube eligible patient was replaced with a modified EAdi catheter. Then the patients were switched to a Servo-i ventilator. According to a random digits table, eligible patients were allocated randomly to ventilation with NAVA or pressure support ventilation (PSV). In PSV group, ventilator settings were determined by the physicians who in charge of the patients, and EAdi signals were not available for ventilator settings. In NAVA group, a daily NAVA level titration was performed to select the NAVA level which got approximate 50% unload, if the patients can't tolerate PSV or NAVA, PCV should be used to insure the ventilation safety. If the patients were under PCV mode, screening should be done by the researchers every 3 hours to make sure whether they will tolerate PSV or NAVA. In both group, daily measurement of diaphragmatic function was performed (only preformed in the first 10 patients of each group), followed by a 30 minutes SBT with PSV 5-7 cmH2O. Patients who were able to tolerate the SBT were extubated. Patients who completed the SBT and remained extubated > 48 h were considered successfully extubated. Patients who failed SBT, or required noninvasive ventilation (NIV), or were re-intubated, or deceased within 48h post-extubation were considered extubation failure. Local sedation protocol including daily wakeup was performed during the research period. All continuous sedative infusions were discontinued at least 1 hour before the measurement of diaphragmatic function and SBT. Main end point was the duration of weaning, and second end point was extubation rate, diaphragmatic function and patient ventilator asynchrony.

ELIGIBILITY:
Inclusion Criteria:

Intubated patients who were deemed ready for weaning by the clinical team but failed the first spontaneous breathing trials (SBT) or weaning

Exclusion Criteria:

1. age <18 or >80 years,
2. tracheostomy
3. treatment abandonment
4. history of esophageal varices
5. gastro-esophageal surgery in the previous 12 months or gastro-esophageal bleeding in the previous 30 days
6. coagulation disorders (INR ratio>1.5 and APTT>44 s)
7. history of acute central or peripheral nervous system disorder or severe neuromuscular disease
8. history of leukemia, severe chronic liver or chronic cardiac disease
9. solid organ transplantation
10. malignant tumor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Duration of weaning | 48h after extubation
  Duration of weaning was defined as time from study enrollment to extubation.

SECONDARY OUTCOMES:
Extubation rate | 48h after extubation or 30 day after enrollment
  Extubation rate was defined as the percentage of patients with successful weaning
diaphragmatic function | At 8 am daily before extubatiuon
  Diaphragmatic function was measured by neuro-ventilatory efficiency (NVE), a ratio of tidal volume to diaphragm electrical activity (Vt/EAdi), and neuro-mechanical efficiency (NME), a ratio of airway pressure to EAdi(Paw/EAdi) during airway occlusion. diaphragmatic function
Patient ventilator asynchrony | At 8 am daily until extubation
  Time delay between neuro inspiration and ventilator delivery. Time delay between neuro expiration and ventilator cycle-off.

OTHER OUTCOMES:
Mortality | ICU or hospital discharge or 28day
  ICU, 28 day and hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, PhD,MD, Study Director — Southeast University
Locations (1):
- Nanjing Zhong-Da Hospital, Nanjing, Jiangsu, China